CLINICAL TRIAL: NCT02183129
Title: Open Label Study to Assess the Efficacy and Safety of Meloxicam 7.5mg vs. Diclofenac 100mg SR in Patients With Osteoarthritis of the Knee
Brief Title: Study to Assess the Efficacy and Safety of Meloxicam vs. Diclofenac SR in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107.229
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Diclofenac; Meloxicam

ARMS (2):
- Meloxicam (Experimental)
  Interventions: Drug: Meloxicam
- Diclofenac (Active Comparator)
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Diclofenac
  Arms: Diclofenac
Drug: Meloxicam
  Arms: Meloxicam

SUMMARY:
To assess the efficacy and safety of meloxicam 7.5mg once daily compared with diclofenac 100mg SR once daily over a treatment period of 8 weeks

ELIGIBILITY:
Inclusion Criteria:

- Osteoarthritis of the knee requiring the therapy with non-steroidal anti-inflammatory drugs (NSAIDs)

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 1999-04-01 (Actual); Primary Completion 1999-11-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain on active movement assessed by a 100 mm visual analogue Scale (VAS) | Baseline, 8 weeks after first drug administration

SECONDARY OUTCOMES:
Change from baseline in Lequesne index | Baseline, 8 weeks after first drug administration
Change from baseline in global assessment by the patient and doctor on a 3-point scale | Baseline, 8 weeks after first drug administration
Number of patients with significant changes from baseline in Laboratory values | Baseline, 8 weeks after first drug administration
Number of patients with significant changes from baseline in physical examinations | Baseline, 8 weeks after first drug administration
Number of patients with Adverse Events | Up to 8 weeks after first drug administration